CLINICAL TRIAL: NCT04377711
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Ciclesonide Metered-Dose Inhaler in Non-hospitalized Patients 12 Years of Age and Older With Symptomatic COVID-19 Infection
Brief Title: A Study of the Safety and Efficacy of Ciclesonide in the Treatment of Non-hospitalized COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Covis Pharma S.à.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALV-020-001
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Results first posted 2022-01-06 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Participants receive Alvesco 320mcg, twice daily for 30 days via pMDI
  Interventions: Drug: Ciclesonide
- Group 2 (Placebo Comparator): Participants receive Placebo matching Alvesco , twice daily for 30 days via pMDI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — 160mcg Inhaler
  Other Names: Alvesco
  Arms: Group 1
Drug: Placebo — Matching Placebo Inhaler
  Arms: Group 2

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Alvesco (ciclesonide) Inhalation Aerosol in non hospitalized patients with symptomatic COVID-19 infection in a multicenter, randomized, double-blind, placebo controlled study

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, efficacy, and safety study of ciclesonide MDI for the treatment of symptomatic COVID-19 infection. Enrolled patients were male and female adults and adolescents 12 years of age or older with confirmed COVID-19 infection who were currently exhibiting symptoms of the disease and who were not currently hospitalized or under immediate consideration for hospitalization at the time of enrollment. The study consisted of an initial screening/enrollment/randomization visit, a 30-day treatment period, and a follow-up period.

ELIGIBILITY:
Inclusion Criteria

Patients eligible for enrollment in the study must meet all the following criteria:

1. Male and female adults and adolescents (12 years of age and above).
2. Positive SARS-CoV-2 rapid molecular diagnostic test within 72 hours prior to enrollment.
3. Patient is not currently hospitalized or under immediate consideration for hospitalization at the time of enrollment.
4. Patient is currently experiencing symptoms of fever, cough, and/or dyspnea.
5. Patient has an oxygen saturation level greater than 93%.
6. Ability to show adequate use of MDI, including inhalation technique.
7. Patient, parent/legal guardian, or legally-authorized representative must have signed a written informed consent before administration of any study-specific procedures.

Exclusion Criteria

Patients meeting any of the following criteria are not eligible for participation in the study:

1. Existence of any life-threatening co-morbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion.
2. History of hypersensitivity to ciclesonide.
3. Treatment with inhaled or intranasal corticosteroids within 14 days of the screening/ enrollment/randomization visit.
4. Treatment with oral corticosteroids within 90 days of the screening/enrollment/randomization visit.
5. Participation in any other clinical trial or use of any investigational agent within 30 days of the screening/enrollment/randomization visit.
6. Currently receiving treatment with hydroxychloroquine/chloroquine.
7. Patients with cystic fibrosis.
8. Patients with idiopathic pulmonary fibrosis.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemency BM, Varughese R, Gonzalez-Rojas Y, Morse CG, Phipatanakul W, Koster DJ, Blaiss MS. Efficacy of Inhaled Ciclesonide for Outpatient Treatment of Adolescents and Adults With Symptomatic COVID-19: A Randomized Clinical Trial. JAMA Intern Med. 2022 Jan 1;182(1):42-49. doi: 10.1001/jamainternmed.2021.6759. PMID 34807241
- [Derived] Farne H, Singanayagam A. Reply. J Allergy Clin Immunol. 2021 Mar;147(3):1117-1118. doi: 10.1016/j.jaci.2020.11.019. Epub 2020 Dec 30. No abstract available. PMID 33388170
- [Derived] Nicolau DV, Bafadhel M. Inhaled corticosteroids in virus pandemics: a treatment for COVID-19? Lancet Respir Med. 2020 Sep;8(9):846-847. doi: 10.1016/S2213-2600(20)30314-3. Epub 2020 Jul 30. No abstract available. PMID 32738928

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciclesonide Arm: Participants receive Alvesco 320mcg, twice daily for 30 days via pMDI
  Ciclesonide: 160mcg Inhaler
- Placebo Arm: Participants receive Placebo matching Alvesco , twice daily for 30 days via pMDI
  Placebo: Matching Placebo Inhaler
Period: Overall Study
Arm/Group | Ciclesonide Arm | Placebo Arm
Started | 197 | 203
Completed | 178 | 181
Not Completed | 19 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 197 | 203 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (17.53) | 42.9 (16.28) | 43.3 (16.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 109 | 221
  Male | 85 | 94 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 86 | 172
  Not Hispanic or Latino | 111 | 117 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 20 | 27 | 47
  White | 174 | 171 | 345
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of COVID-19-related Symptoms by Day 30
Description: Time to alleviation of COVID-19-related symptoms of cough, dyspnea, chills, feeling feverish, repeated shaking with chills, muscle pain, headache, sore throat, and new loss of taste or smell, defined as symptom-free for a continuous period of more than 24 hours (ie, later than 3 AM/PM assessments) by day 30
Time Frame: Day 30
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ciclesonide Arm | Placebo Arm
Number analyzed (Participants) | 197 | 203
days | 19.0 [14.0 to 21.0] | 19.0 [16.0 to 23.0]

2. Secondary Outcome: Percentage of Patients With Hospital Admission or Death by Day 30
Description: Assess whether treatment with ciclesonide MDI (Metered Dose Inhaler) plus standard supportive care reduces the incidence of hospital admissions or death compared with placebo plus standard supportive care in non-hospitalized patients with symptomatic COVID-19 infection.
Time Frame: Day 30
Measure: Number; unit: percentage of patients
Arm/Group | Ciclesonide Arm | Placebo Arm
Number analyzed (Participants) | 197 | 203
percentage of patients | 1.5 | 3.4

3. Secondary Outcome: All-cause Mortality by Day 30
Description: Assess whether treatment with ciclesonide MDI plus standard supportive care reduces all-cause mortality compared with placebo plus standard supportive care in non-hospitalized patients with symptomatic COVID-19 infection.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Arm | Placebo Arm
Number analyzed (Participants) | 197 | 203
Participants | 0 | 0

4. Secondary Outcome: COVID-19-related Mortality by Day 30
Description: Assess whether treatment with ciclesonide MDI plus standard supportive care reduces COVID-19-related mortality compared with placebo plus standard supportive care in non-hospitalized patients with symptomatic COVID-19 infection.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Arm | Placebo Arm
Number analyzed (Participants) | 197 | 203
Participants | 0 | 0

5. Secondary Outcome: Percentage of Patients With Subsequent Emergency Department Visit or Hospital Admission for Reasons Attributable to COVID-19 by Day 30
Description: Assess whether treatment with ciclesonide MDI plus standard supportive care reduces the incidence of subsequent emergency department visits or hospital admissions for reasons attributable to COVID-19 compared with placebo plus standard supportive care in non-hospitalized patients with symptomatic COVID-19 infection
Time Frame: Day 30
Measure: Number; unit: percentage of patients
Arm/Group | Ciclesonide Arm | Placebo Arm
Number analyzed (Participants) | 197 | 203
percentage of patients | 1.0 | 5.4

6. Secondary Outcome: Percentage of Patients With Alleviation of COVID-19-related Symptoms Defined as Symptom-free for a Continuous Period of More Than 24 Hours (ie, Later Than 3 AM/PM Assessments) by Day 7, by Day 14, and by Day 30
Description: Assess whether treatment with ciclesonide MDI plus standard supportive care increases the percentage of patients with alleviation of COVID 19-related symptoms of cough, dyspnea, chills, feeling feverish, repeated shaking with chills, muscle pain, headache, sore throat, and new loss of taste or smell compared with placebo plus standard supportive care in non-hospitalized patients with symptomatic COVID-19 infection.
Time Frame: By day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Ciclesonide Arm | Placebo Arm
Number analyzed (Participants) | 197 | 203
Participants | 139 | 129

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 30-day treatment period and 60-day follow up period.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/203
Serious Adverse Events (participants affected / at risk) | 3/197 | 7/203
Other Adverse Events (participants affected / at risk) | 22/197 | 29/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=197) | Group 2 (N=203)
COVID-19, renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oxygen saturation decreased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation, COVID-19 pneumonia (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 (i.e., worsening of COVID-19) (Infections and infestations) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=197) | Group 2 (N=203)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Headache (General disorders) | 1 | 4
Dry Mouth (Gastrointestinal disorders) | 3 | 1
COVID-19 (ie, worsening of COVID-19 (Infections and infestations) | 1 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 2
Oral Candidiasis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Piriformis syndrome (Nervous system disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT04377711/Prot_SAP_000.pdf